CLINICAL TRIAL: NCT02804217
Title: Identification of Genomic Mutation Profile Using Next Generation Sequencing for Non-small-cell Lung Cancer Patients With Activating EGFR Mutations Harboring Acquired Resistance to the First-generation EGFR TKIs.
Brief Title: Acquired Resistant Mechanism of the First-generation EGFR TKIs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yu Xinmin, Director, Zhejiang Cancer Hospital
Other Study IDs: IRB-2016-74
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Non-small Cell Lung Cancer; Aquired Resistance; EGFR TKIs
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Genetic: mutation profile
  Other Names: Procedure: Lung tumor biopsy; Procedure: Blood sample

SUMMARY:
Patients with advanced non-small-cell lung cancer (NSCLC) harboring sensitive epithelial growth factor receptor (EGFR) mutations invariably develop acquired resistance to EGFR tyrosine kinase inhibitors (TKIs). Identification of actionable genetic mutations can be helpful for guiding the subsequent treatment. This study aimed to analyze the genetic profile of NSCLC harboring acquired resistance to the first-generation EGFR TKIs using next generation sequencing (NGS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage IIIB or IV non-small cell lung cancer
* patients harboring sensitive EGFR mutations and received first-generation EGFR-TKIs who developed acquired drug resistance
* patients who can provide pre-treatment (EGFR TKIs) tumor tissues
* patients with tumor lesions to be re-biopsy after drug resistance
* patients must sign an informed consent indicating that they are aware of the .investigational nature of the study in keeping with the policy of the hospital.

Exclusion Criteria:

* History of another malignancy except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* patients with other systemic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with NSCLC harboring sensitive EGFR mutations and received first-generation EGFR-TKIs who developed acquired drug resistance
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
mutation profile | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China